CLINICAL TRIAL: NCT00658944
Title: Preoperative MUCP and VLPP Failed to Predict Long Term (4-Years) Outcome in Patients Who Underwent Transobturator Mid-Urethral Slings. a Prospective Observational Descriptive Study
Brief Title: Predictive Objective Parameters for Outcome of the Treatment of Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Elisabetta Costantini, Department of Medical-Surgical Specialties, Section of Urology and Andrology
Other Study IDs: EC_ML_002; EC_ML_002s
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Urinary Incontinence
Keywords: Stress urinary incontinence; Mixed urinary incontinence; surgery; trans obturator tape; Maximum urethral closure pressure; Valsalva leak point pressure; outcome
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients suffering from stress or mixed urinary incontinence

SUMMARY:
To investigate the role of preoperative maximum urethral closure pressure and Valsalva leak point pressure in predicting outcome in patients who underwent trans-obturator tape for the treatment of female stress urinary incontinence.

DETAILED DESCRIPTION:
A prospective observational descriptive study conducted from May 2002 to November 2005 at a single tertiary urban teaching University Uro-gynecological Department. 65 patients affected by stress or mixed urinary incontinence (stress component clinically predominant), defined according to International Continence Society guidelines, associated or not with urethral hypermobility underwent surgery which consisted of a fusion-welded, non-woven, non-knitted polypropylene tape (Obtape® Mentor-Porges). Preoperative MUCP and VLPP, stratified as ≤ or > 40 cmH20 and ≤ or > 60 cmH2O respectively, were separately or in combination correlated with primary (continence status: dry or wet) and secondary outcome variables (QoL questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Mixed urinary incontinence (stress component clinically predominant)

Exclusion Criteria:

* > grade II uro-genital prolapse in any vaginal compartment
* Previous incontinence surgery
* Urine retention, neurogenic bladder, benign or malignant uterus lesion (leiomyoma, fibromyoma, cervical or endometrial carcinoma)
* Active pelvic inflammatory disease
* Known hypersensitivity to synthetic materials (polypropylene, polythetrafloroethilene, polyethileneterephtalate, polyglactil acid or polyglycolic acid)
* Pregnancy or lactation; AND
* Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stress or mixed urinary incontinence (stress component clinically predominant), defined according to ICS guidelines, associated or not with urethral hypermobility
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2002-05; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Costantini, MD, Principal Investigator — University Of Perugia
Locations (1):
- Department of Urology, Perugia, Perugia, Italy

REFERENCES:
- See also: Web site of University of Perugia — http://www.unipg.it